CLINICAL TRIAL: NCT06206304
Title: Evaluation of the Relationship Between Eye Color and Post-Operative Pain in Female Patients Experiencing Symptomatic Irreversible Pulpitis in A Mandibular Molar: A Prospective, Parallel-Group, Observational Clinical Study
Brief Title: Relationship of Eye Colour With Anesthetic Success and Post-Operative Pain
Status: Completed | Type: Observational
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Merve Sari, Assistant Professor, Mustafa Kemal University
Other Study IDs: 231412
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Post-operative Pain; Irreversible Pulpitis
Keywords: eye color; inferior alveolar nerve block; irreversible pulpitis; phenotype; post-operative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Root Canal Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Light-eyed females: Blue-green colors were categorized as light
  Interventions: Other: Root canal therapy
- Dark-eyed females: All shades of brown were categorized as dark.
  Interventions: Other: Root canal therapy

INTERVENTIONS:
Other: Root canal therapy — Traditional root canal therapy was performed with rubber-dam isolation.

SUMMARY:
Current evidence indicates that some phenotypic characteristics, such as eye or hair color, might be associated with the experience of pain. We therefore compared the anaesthetic success rate of inferior alveolar nerve block (IANB), and post-operative pain scores between light and dark eyed in female patients experiencing symptomatic irreversible pulpitis (SIP) in a mandibular molar.

110 adult patients, experiencing moderate or severe pain with SIP, participated in this prospective study. All patients received IANB of 4% articaine with 1:100.000 epinephrine. Endodontic access cavity preparation was initiated after confirmed of IANB with numbness of the lower lip. Pain during treatment was recorded by using a Heft Parker Visual Analog Scale. Anaesthetic success was recorded as ''none'' or ''mild'' pain. Root canal treatment was performed, with standardized protocols. Post-operative pain scores were also recorded 24, 48, 72 hours and 7 days after treatment.

DETAILED DESCRIPTION:
Female patients with no systemic diseases (ASA 1-2); aged between 18-45 years; eye colors with brown, hazel, green, or blue; mandibular molar teeth diagnosed SIP were included in this study.

Categorization Of The Patient's Eye Color Categorization of the patient's eye color was made by an independent researcher. Patients were also asked to indicate their own eye color. If a consensus could not be reached between the researcher and the patient regarding eye color, the patient was excluded from the study. Blue-green colors were categorized as light; all shades of brown were categorized as dark.

Root Canal Treatment Procedures All dental procedures, including anesthesia injection, were performed by a single endodontist. 119 patients received IANB injections of 1.8 mL 4% articaine with 1:100,000 epinephrine (Ultracain D-S; Sanofi, Paris, France) using Halstead method. 27-gauge needle (Beybi Medical Co., Istanbul, Turkey) were used for all injections. Anesthetic solution was slowly deposited to the target area for 60 seconds. 10 minutes after IANB anesthesia, patients were asked whether their lip were numb. Patients who reported no profound lip numbness were excluded from the study. An access cavity was prepared using a high speed steril diamond bur #801G (Meisinger) under abundant water coolant after isolation with a rubber dam. Patients were instructed to inform the operator if they felt pain during acces cavity preparation. Pain intensity was rated into 4 categories using the HP VAS.

Level 1: No pain (0) Level 2: Mild pain (1-3 mm) Level 3: Moderate pain (4-6mm) Level 4: Severe pain (7-10 mm). The IANB anesthesia was defined as successful when the patient reported no pain or mild pain during cavity preparation. The IANB anesthesia was considered unsuccessful in patients with moderate or severe pain; in these cases, an intrapulpal anesthesia was performed.

After localizing the canal orifices, the working length (WL) was determined using a 10 K file (VDW, Munich, Germany), to be 0.5 mm shorter than the "0.0" reading on the apex locator (Morita Root ZX, Japan), and confirmed by radiographs. Root canal were prepared using the R25 (Reciproc, VDW) file in the mesial root canals and the R25, R40, and R50 files in the distal root canals, respectively, with crown-down technique. After 3 pecking motions the file was removed from the root canal and debris on the file surface was cleaned. The pecking depth for the pecking motions were 3-4 mm. Each root canals was irrigated a total of 20 ml of 2,5% sodium hypochlorite (NaOCl; Wizard, RehberKimya, Istanbul, Turkey) solution using 30 G irrigation needle (Medic; Shangai Carelife, China). After NaOCl. 5 ml of distilled water used to neutralize the effect of NaOCl. The final irrigation was performed with 3 mL 17% ethylenediaminetetraacetic acid (EDTA; Coltene, Altstatten, Switzerland) solution. The Endoactivator (EA; Dentsply Tulsa Dental Specialties, Tulsa, OK) 25/04 tip placed 2 mm behind the WL was used in 3 cycles of 20 s each. EDTA was activated with 2-4 mm vertical movements for 1 min using the EA. 5 ml of distilled water used to neutralize the effect of EDTA followed by the root canals were dried with paper points (VDW). The root canals were filled with the lateral condensation using gutta-percha cones (VDW) and epoxy-resin-based sealer (AH Plus; Dentsply DeTrey GmbH, Konstanz, Germany) in a single visit. All teeth were restored with resin composite (Estelıte Sıgma Quıck; Tokuyama, Tokyo, Japan). The root canal filling was checked by radiographs.

If any complications such as broken file, ledging, could not be reached to the WL; overfilling (filling beyond the radiographic apex) or short filling (>2 mm from the radiographic apex) the patient was excluded from the study.

The patients were prescribed 400 mg of ibuprofen, and instructed to take it only in the presence of pain. Patients were asked to rate their post-op pain on the HP VAS scale at hours 24h, 48 h, 72h and on day 7 after the treatment and to record analgesic drugs they used.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no systemic diseases
* Eye colors with brown, hazel, green, or blue; mandibular molar teeth diagnosed with SIP The diagnosis of SIP was confirmed by a a prolonged response to cold test (Endo Ice; Coltene, Altstatten, Switzerland) and positive response to electric pulp testing. Only patients with moderate (4-6 mm) or severe pain (7-10 mm) according to HP VAS were included.
* Teeth with no periodontal problem (probing pocket depth ≤3 mm and mobility within normal limit) and without periapical radiolucency (except for a widened periodontal ligament with an intact lamina dura) were included.

Exclusion Criteria:

- Patients using colored contact lenses; any surgical operation to change iris color; neurophysiological disease; taking any medications that may affect pain or anxiety assessment (nonsteroidal anti-inflammatory drugs, opioids, antidepressants, and alcohol), pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility was based on self-representation of gender identity
Study Population: University endodontics clinic
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-06-18 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
post-operative pain | 1 week
  Pre-operative and post-operative pain scores were determined according to the Heft-Parker Visual Analog Scale (HP VAS), which consisted of a 10 mm long horizontal line where numerical values were divided into visual categories.
  Patients were instructed to score their pain with a value on the HP VAS. The presence or absence of pain was classified according to 4 categories: No pain (level 1, 0), Mild pain (level 2, 1-3 mm), Moderate pain (level 3, 4-6mm), Severe pain (level 4, 7-10 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Merve Sarı, DDS, Principal Investigator — Mustafa Kemal University; Koray Yılmaz, DDS,MSc, Study Director — Cukurova University
Locations (2):
- Turkey (Türkiye) (2):
  - Department of Endodontics, Faculty of Dentistry, Hatay Mustafa Kemal University, Hatay, Antakya
  - Mustafa Kemal University, Hatay, Antakya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Droll B, Drum M, Nusstein J, Reader A, Beck M. Anesthetic efficacy of the inferior alveolar nerve block in red-haired women. J Endod. 2012 Dec;38(12):1564-9. doi: 10.1016/j.joen.2012.08.014. Epub 2012 Oct 3. PMID 23146638
- [Background] Liem EB, Joiner TV, Tsueda K, Sessler DI. Increased sensitivity to thermal pain and reduced subcutaneous lidocaine efficacy in redheads. Anesthesiology. 2005 Mar;102(3):509-14. doi: 10.1097/00000542-200503000-00006. PMID 15731586
- [Background] SUTTON PR. Association between colour of the iris of the eye and reaction to dental pain. Nature. 1959 Jul 11;184:122. doi: 10.1038/184122a0. No abstract available. PMID 13835852
- [Background] Hyde J, Fowler S, Drum M, Reader A, Nusstein J, Beck M. Is Eye Color Related to Dental Injection Pain? A Prospective, Randomized, Single-blind Study. J Endod. 2018 May;44(5):734-737. doi: 10.1016/j.joen.2018.01.009. Epub 2018 Mar 2. PMID 29506886
- [Background] Mogil JS, Wilson SG, Chesler EJ, Rankin AL, Nemmani KV, Lariviere WR, Groce MK, Wallace MR, Kaplan L, Staud R, Ness TJ, Glover TL, Stankova M, Mayorov A, Hruby VJ, Grisel JE, Fillingim RB. The melanocortin-1 receptor gene mediates female-specific mechanisms of analgesia in mice and humans. Proc Natl Acad Sci U S A. 2003 Apr 15;100(8):4867-72. doi: 10.1073/pnas.0730053100. Epub 2003 Mar 27. PMID 12663858
- [Background] Liem EB, Lin CM, Suleman MI, Doufas AG, Gregg RG, Veauthier JM, Loyd G, Sessler DI. Anesthetic requirement is increased in redheads. Anesthesiology. 2004 Aug;101(2):279-83. doi: 10.1097/00000542-200408000-00006. PMID 15277908
- [Derived] Sari M, Yilmaz K. Association Between Eye Color and Postoperative Pain in Female Patients With Symptomatic Irreversible Pulpitis in Mandibular Molars: A Prospective, Parallel-Group, Observational Study. Pain Res Manag. 2024 Oct 23;2024:8824366. doi: 10.1155/2024/8824366. eCollection 2024. PMID 39479199